CLINICAL TRIAL: NCT03558269
Title: Pilot Study to Assess the Efficacy of Autologous Umbilical Cord Blood Treatment of Brain and Heart Injury in Neonates With Congenital Heart Defect
Brief Title: Autologous Umbilical Cord Blood Treatment of Neonate With CHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Omer Bar-Yosef, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3757-16-SMC
Record Dates: First submitted 2018-05-12; First posted 2018-06-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Congenital Heart Disease; Brain Injuries; Low Cardiac Output Syndrome; Neonatal Disorder
Keywords: Autologous Umbilical cord blood infusion; Congenital Heart Disease; Brain Injuries; Low Cardiac Output Syndrome; Neonatal Disorder
MeSH Terms: conditions — Heart Defects, Congenital; Brain Injuries; Cardiac Output, Low; Infant, Newborn, Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be exposed to the participant group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group will receive UCB after the first palliative surgery
  Interventions: Biological: Autlogous UCB infusion
- Control group (No Intervention): This group will not receive any treatment

INTERVENTIONS:
Biological: Autlogous UCB infusion — Infants delivered with hypoplastic left heart syndrome and transposition of great arteries undergoing surgery in the 1st 2 weeks of life will be treated with autologous UCB after the surgery. Each group will be followed by MRI before (1-3 days) and after the surgery between at 10 POD. Developmental follow up will be done at 1, 6 and 12 months. Another brain MRI will be done at 6 months of age.
  Arms: Study group

SUMMARY:
The aim of the study is to evaluate the feasibility and safety and efficacy of collecting and infusing autologous umbilical cord blood (UCB) in newborn infants with hypoplastic left heart syndrome (HLHS) and transposition of great arteries (TGA).

Rationale: Neonates with HLHS and TGA have significant brain injury as demonstrated by peri-surgical MRI. Moreover, there a substantial tendency to suffer from chronic cardiac condition as low cardiac output state and valvular insufficiency. Treatment of neonates after hypoxic ischemic injury at birth with autologous UCB was shown to safe and improved developmental outcome. The effect of UCB is most likely achieved by reduction of free radicals injury and pro-inflammatory and apoptotic process.

Hypothesis: Treatment with UCB immediately after the first cardiac surgey, with in the first week life will reduce the brain injury demonstrated by MRI and reduce the choronic cardiac problems

DETAILED DESCRIPTION:
The aim of this pilot study is to evaluate the safety and feasibility of infusion of autologous umbilical cord blood (UCB) in neonates with with hypoplastic left heart syndrome (HLHS) or transposition of great arteries (TGA).

This is a prospective, matched control study, Phase I-II trial to evaluate the safety and efficacy of autologous UCB infusion in neonates with HLHS or TGA. The study group will consist of neonate that were diagnosed by prenatal fetal ultrasound with HLHS or TGA and their UCB was collected at the time of delivery.

The study group will include the patients with UCB and the control group will be patients without UCB.

All patients will have their surgery within 2 weeks from birth. The UCB will be infused to the patients in study group as soon as the patient has stabilized after the surgery and not more than 7 days after surgery.

Both groups will be followed similarity:

During hospitalization:

Neurological and cardiac evaluation a day before surgery, 7 days after surgery and at discharge.

Blood tests for immune and growth factors a day before surgery, at the time of infusion (or intended infusion for the control group) ,1 and 7 days after infusion.

have a cardiac and brain MRI before the surgery and within 14 days after surgery.

Brain and cardiac MRI before surgery, 7-14 days after surgery.

Ambulatory follow up (similar to routine follow up):

Cardiac and neuro-developmental evaluation at 1,6,12 month Blood tests for immune and growth factors at 1 month

ELIGIBILITY:
Inclusion Criteria:

1. At least 35 weeks of gestation
2. Prenatal diagnosis of HLHS including mitral stenosis/atresia, aortic stenosis/atresia, arch hypoplasia and the presence of hypoplastic left ventricle with or without VSD.
3. Norwood procedure will take place within 14 days from birth.
4. Treatment with cord blood should be given within 7 days after surgery.
5. Parental informed consent for collection of umbilical cord blood.

Exclusion Criteria:

1. Total nucleated cells (TNC) lower than 1X107 in the collected umbilical cord blood unit.
2. Infected umbilical cord blood unit.
3. Parents refusal to continue in the study at any stage.

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging of the brain before and after the surgery (ref 1) | The time frame between MRI before and after surgery is 10-13 days
  Change in MRI of the brain before (between 1-3 days) and after (10 days) the surgery between the intervention and control group. The change will be quantified by MRI brain injury severity (BIS) score quantifying white matter injury, stroke and brain hemorrhage. Diffusion tensor imaging measures will also be quantified by using average diffusivity and fractional anisotropy calculated from frontal, parietal, temporal and occipital white matter.

SECONDARY OUTCOMES:
Neuro-development at one month | One month
  General movements assessment (ref 2)
Neuro-development at six month | 6 months
  Gross Motor Function Measure 66 (ref 3)
Neuro-development at 12 month | 12months
  Gross Motor Function Measure 66 (ref 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
By excel data base

REFERENCES:
- [Background] Kwong AKL, Fitzgerald TL, Doyle LW, Cheong JLY, Spittle AJ. Predictive validity of spontaneous early infant movement for later cerebral palsy: a systematic review. Dev Med Child Neurol. 2018 May;60(5):480-489. doi: 10.1111/dmcn.13697. Epub 2018 Feb 22. PMID 29468662
- [Background] Alotaibi M, Long T, Kennedy E, Bavishi S. The efficacy of GMFM-88 and GMFM-66 to detect changes in gross motor function in children with cerebral palsy (CP): a literature review. Disabil Rehabil. 2014;36(8):617-27. doi: 10.3109/09638288.2013.805820. Epub 2013 Jun 26. PMID 23802141
- [Result] Dimitropoulos A, McQuillen PS, Sethi V, Moosa A, Chau V, Xu D, Brant R, Azakie A, Campbell A, Barkovich AJ, Poskitt KJ, Miller SP. Brain injury and development in newborns with critical congenital heart disease. Neurology. 2013 Jul 16;81(3):241-8. doi: 10.1212/WNL.0b013e31829bfdcf. Epub 2013 Jun 14. PMID 23771484